CLINICAL TRIAL: NCT03611426
Title: A Randomized，Ascending Dose，Single-blind Phase 1&2 Study to Evaluate the Safety, Tolerability, Immunogenicity and Efficacy of Topical rhThrombin as an Adjunct to Hemostasis During Segmental Hepatectomy
Brief Title: Topical rhThrombin as an Adjunct to Hemostasis During Segmental Hepatectomy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: ZGrhT001
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2019-10

CONDITIONS: Hepatectomy
Keywords: Serine protease; Tolerance; Immunogenicity; Safety
MeSH Terms: interventions — recombinant human thrombin

STUDY DESIGN:
Intervention Model Description: The first part is ascending dose study: 3 subjects take rhThromb and 1 subjects take the same volume of saline; The second part is dose extension study:2 cohorts and 1 blank control group( the same volume of saline) used with absorbable collagen sponge;every group need 12 subject; The second part is dose extension study: 2 cohorts and 1 blank control group( the same volume of saline);every group need 12 subject;
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhThrombin ( Topical ) (Experimental): Cohort 1:rhThrombin ( Topical ) 500IU /ml、1000IU/m and 2000IU/ml During segmental hepatectomy; Cohort 2:rhThrombin ( Topical ) 1000IU/m and 2000IU/ml with absorbable collagen sponge During segmental hepatectomy; Cohort 3:rhThrombin ( Topical ) 1000IU/m and 2000IU/ml used directly sprayed on hemorrhagic point During segmental hepatectomy;
  Interventions: Drug: rhThrombin ( Topical )
- placebo (Placebo Comparator): Cohort 1: the same volume of saline during segmental hepatectomy; Cohort 2:the same volume of saline used withabsorbable collagen sponge during segmental hepatectomy; Cohort 3:the same volume of saline during segmental hepatectomy;
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rhThrombin ( Topical ) — Active Substance
  Other Names: Recombinant Human Thrombin (CHO Cell) for Topical Use
  Arms: rhThrombin ( Topical )
Drug: placebo — saline solution
  Other Names: PLA
  Arms: placebo

SUMMARY:
rhThrombin is a serine protease from human.The study is to assess the Safety, Tolerability, Immunogenicity and efficacy of rhThrombin.

DETAILED DESCRIPTION:
The study is a randomized, single-blind,blank controlled phase 1&2 trial ,including 3 independent parts toevaluate the safety,efficacy and immunogenicity.

The first part is ascending dose,blank control tolerability and safety study. The Starting doses from 500IU/ml to 1000IU/mL and 2000IU/mL to evaluate the safety,efficacy.

The second part is randomized, single-blind, blank controlled study to evaluate safety、efficacy and immunogenicity. Doses settings :1000IU/mL , 2000IU/mL and blank group which with absorbable collagen sponge when used.

The third part is randomized, single-blind, blank controlled study to evaluate safety、efficacy and immunogenicity. Doses settings :1000IU/mL , 2000IU/mL and blank group which directly sprayed on hemorrhagic point when used.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 18 and 75 years of age;
2. Hepar wedge resection or anatomic hepatectomy(one to five continue hepatic segments) (remark:including open surgery or hand-assisted laparoscopic surgery,patients who has been cholecystectomy or choledochotomy can be also get into the study);
3. Blood routine(including WBC、ANC、RBC、Hb and PLT) and Liver function(ALT≤1.5ULN、AST≤1.5ULN) is appear normal. ALP、LDH、 TBil、Dbil are normal.(Remark: Patients whose Laboratory tests are abnormal but they are no clinical significance can get into the study);
4. Renal function(including Cr、BUN)、coagulation function（including PT、APTT、TT、INR）、 electrolytes（include K、Na、CL、Ca、P、Mg）and electrocardiogram are normal or anormal.Investigator think they make no difference to operation;
5. No other therapeutic surgery was performed in the first 4 weeks before the subject gets into clinical research the study(in addition to diagnostic surgery).
6. Patients have not used blood products in 24hours before surgery.
7. Meet the requirements of the ethics committee.Sign the informed consent form and visited according to the protocol.

Exclusion Criteria:

1. Blood system diseases are known, including coagulopathy or bleeding tendency;
2. Life signs were not stable for more than 24hours;
3. Severe heart、brain and blood vessel diseases in past 6 months,including TIA、Non-disabling cerebral infarction、myocardial infarction、unstable angina or Intracranial hemorrhage;
4. Using the drugs that have an effect on blood coagulation in 7 days before surgey(including but not limited to: aspirin、clopidogrel、ticlopidine、dipyridamole、ginkgo biloba extract、heparin、warfarin、citrates、hemocoagulase、VitK、ethamsylate and Vitc,etc);
5. Complicated with other serious diseases(active infections,uncontrolled diabetes and hyperthyroidism);
6. Be allergic to thrombin(human)、serum(snake) and proteins (hamster);
7. Female subjects are in lactation or serum pregnancy test are positive;
8. Take part in other clinical trail within 4 weeks before geting into the study;
9. Using the Thrombin products and Antithrombin antibodies or Coagulation V factor antibodies are positive before, after using rhthrombin, it may generate an immune response.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of adverse events | baseline to 4 weeks
  Incidence and Severity of adverse events

SECONDARY OUTCOMES:
Proportion of Subjects Achieving Hemostasis by Six Minutes After Treatment Start | From start of treatment until 6 minutes after treatment start
  Subjects achieving hemostasis at the target bleeding site by 6 minutes following the start of treatment without the occurrence of re-bleeding until the completion of surgical closure
The hemostatic time of the woud | From start of treatment until 6 minutes after treatment start
  The hemostatic time of the woud
immunogenicity | baseline to 4 weeks
  Incidence of rhThrombin antibody and Confirm whether they are neutralizing antibody

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwei Li, PhD, Principal Investigator — The First Affiliated Hospital of Medical School of Zhejiang University
Locations (1):
- Zhiwei Li, Hangzhou, Zhejiang, China